CLINICAL TRIAL: NCT03428217
Title: A Randomized, Double-Blind, Placebo-Controlled Phase 2 Clinical Trial Comparing CB-839 in Combination With Cabozantinib (CB-Cabo) vs. Placebo With Cabozantinib (Pbo-Cabo) in Patients With Advanced or Metastatic Renal Cell Carcinoma (RCC)
Brief Title: CANTATA: CB-839 With Cabozantinib vs. Cabozantinib With Placebo in Patients With Metastatic Renal Cell Carcinoma
Acronym: CANTATA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Calithera Biosciences, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CX-839-008
Record Dates: First submitted 2018-02-05; First posted 2018-02-09 (Actual); Results first posted 2023-03-20 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-02

CONDITIONS: Advanced Renal Cell Carcinoma; Metastatic Renal Cell Carcinoma
Keywords: Tumor Metabolism; RCC; Glutaminase Inhibitor; CB-839; CANTATA; TKI; Tyrosine Kinase Inhibitor; cabozantinib; Cabometyx; Cometriq; glutaminase; glutamine; renal cell; clear cell; kidney cancer; cMET; MET; HGFR; telaglenastat
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms | interventions — CB-839; cabozantinib

STUDY DESIGN:
Intervention Model Description: This is a double blinded placebo-controlled study where patients will be randomized 1:1 to either CB-839 (telaglenastat) plus cabozantinib or placebo plus cabozantinib
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, care providers, investigators and outcomes assessors are blinded to treatment. Progression free survival (PFS) will be assessed by a blinded Independent Radiology Committee for the primary endpoint of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pbo-Cabo (Placebo Comparator): Placebo twice daily (BID) + cabozantinib (60 mg once daily [QD]) administered orally on Days 1 through 28 of each 28-day cycle until disease progression per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) or unacceptable toxicity, whichever occurred first.
  Interventions: Drug: Cabozantinib; Drug: Placebo
- CB-Cabo (Experimental): CB-839 800 mg BID + cabozantinib (60 mg QD) administered orally on Days 1 through 28 of each 28-day cycle until disease progression per RECIST v1.1 or unacceptable toxicity, whichever occurred first.
  Interventions: Drug: CB-839; Drug: Cabozantinib

INTERVENTIONS:
Drug: CB-839 — Oral glutaminase inhibitor
  Other Names: telaglenastat
  Arms: CB-Cabo
Drug: Cabozantinib — Oral receptor tyrosine kinase inhibitor
  Other Names: Cabometyx; Cabometriq
Drug: Placebo — Placebo tablets
  Arms: Pbo-Cabo

SUMMARY:
Tthe primary objective of this study is to compare blinded Independent Radiology Committee (IRC)-adjudicated progression free survival (PFS) of patients treated with CB-839 + cabozantinib (CB-Cabo) versus placebo + cabozantinib (Pbo-Cabo) for advanced or metastatic clear-cell RCC (ccRCC).

ELIGIBILITY:
Inclusion Criteria:

1. Documented histological or cytological diagnosis of renal cell carcinoma with a clear-cell component
2. Adult patients
3. Karnofsky Performance Score (KPS) ≥ 70%
4. Measurable Disease per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1)
5. 1-2 lines of prior therapy for advanced or metastatic renal cell carcinoma (RCC) including one anti-angiogenic therapy (any vascular endothelial growth factor [VEGF] pathway-targeted agent used either as monotherapy or as a component of a combination regimen) OR the combination regimen of nivolumab + ipilimumab
6. Adequate hepatic, renal, cardiac and hematologic function

Exclusion Criteria:

1. Prior treatment with cabozantinib (or other mesenchymal-epithelial transition [MET] inhibitor) or CB-839
2. Receipt of other anticancer therapy within 2-6 weeks, depending on the treatment
3. Untreated or active brain metastases or central nervous system cancer, as defined per protocol
4. Prior gastric surgery, small bowel resection, or other conditions that may impede adequate absorption of oral study drug
5. Known active infection with human immunodeficiency virus (HIV), Hepatitis B or C virus
6. Inability to discontinue proton-pump-inhibitor use before randomization
7. Patients who are pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 444 (Actual)
Dates: Start 2018-04-24 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2021-07-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sam Whiting, M.D., Ph.D., Study Director — Calithera Biosciences, Inc
Locations (133):
- United States (59):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Mayo Clinic Cancer Center, Phoenix, Arizona
  - The University of Arizona Cancer Center, Tucson, Arizona
  - Cedars-Sinai Medical Center, Samuel Oschin Comprehensive Cancer Institute, Los Angeles, California
  - Stanford Cancer Center, Palo Alto, California
  - Salinas Valley Memorial Healthcare System, Salinas, California
  - St. Joseph Heritage Healthcare, Santa Rosa, California
  - Penrose Cancer Center, Research Department, Colorado Springs, Colorado
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Florida Cancer Specialists, Fort Myers, Florida
  - University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida
  - Florida Cancer Specialists, St. Petersburg, Florida
  - H.Lee Moffitt Cancer & Research Institute (Moffitt Cancer Center), Tampa, Florida
  - Emory Winship Cancer Institute, Atlanta, Georgia
  - Georgia Cancer Center at Augusta University, Augusta, Georgia
  - Northwest Georgia Oncology Centers, PC, Marietta, Georgia
  - St. Luke's Mountain States Tumor Institute, Boise, Idaho
  - Northwestern University, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - NorthShore University HealthSystem, Evanston, Illinois
  - AMITA Health Cancer Institute & Outpatient Center, Hinsdale, Illinois
  - Orchard Healthcare Research, Inc., Skokie, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Goshen Center for Cancer Care, Goshen, Indiana
  - East Jefferson General Hospital, Metairie, Louisiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - University of Maryland, Greenebaum Comprehensive Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - HealthPartners Institute, Regions Cancer Care Center, Saint Paul, Minnesota
  - Hattiesburg Clinic Hematology/Oncology, Hattiesburg, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Mercy Hospital, Joplin, Missouri
  - HCA Midwest Health, Kansas City, Missouri
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - San Juan Oncology Associates, PC, Farmington, New Mexico
  - Roswell Park Cancer Center, Buffalo, New York
  - North Shore Hematology Oncology Associates PC dba NY Cancer and Blood Specialists, East Setauket, New York
  - NYU Winthrop Hospital, Mineola, New York
  - Northern Westchester Hospital, Mount Kisco, New York
  - Stony Brook Cancer Center, Stony Brook, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - INTEGRIS Cancer Institute of Oklahoma Proton Campus, Oklahoma City, Oklahoma
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center (UPMC) Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Saint Francis Hospital Cancer Center, Greenville, South Carolina
  - West Cancer Center, Germantown, Tennessee
  - The Sarah Cannon Research Institute, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - The Center for Cancer and Blood Disorders, Fort Worth, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - University of Utah, Huntsman Cancer Institute, Salt Lake City, Utah
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Froedtert Hospital and the Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (14):
  - Southern Highlands Private Hospital (Cancer Centre), Bowral, New South Wales
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - MacQuarie University Hospital, North Ryde, New South Wales
  - Liverpool Hospital, Sydney, New South Wales
  - Tweed Hospital, Tweed Heads, New South Wales
  - Pindara Private Hospital, Benowa, Queensland
  - Cairns Hospital, Cairns, Queensland
  - Mater Misericordiae Limited - Division of Cancer Services, South Brisbane, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Ballarat Health Services, Ballarat, Victoria
  - Peninsula Private Hospital, Frankston, Victoria
  - Cabrini Hospital, Malvern, Victoria
  - Goulburn Valley Health, Shepparton, Victoria
  - Hollywood Private Hospital, Nedlands, Western Australia
- France (16):
  - Centre hospitalier régional universitaire (CHRU) de Besançon - Jean-Minjoz, Besançon
  - CHU de Bordeaux Hôpital Saint André, Bordeaux
  - Centre François Baclesse, Caen
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre hospitalier universitaire (CHU) Henri-Mondor, Créteil
  - Centre Georges-François Leclerc, Dijon
  - Centre Léon Bérard, Lyon
  - Institut Paoli-Calmettes Service d'Urologie, Marseille
  - Institut de Cancérologie de Montpellier (ICM), Montpellier
  - Centre Antoine Lacassagne, Nice
  - Hôpital Européen Georges-Pompidou (HEGP), Paris
  - Institut de Cancérologie de l'Ouest (ICO) - Centre René Gauducheau, Saint-Herblain
  - CHU de Strasbourg (Les Hôpitaux Universitaires de Strasbourg), Strasbourg
  - IUCTO Bureau des Essais Cliniques (Institut Claudius Regaud), Toulouse
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy - Le département de Medecine oncologique, Villejuif
- Germany (7):
  - Medical University Heidelberg, NCT (National Center for Tumour Diseases), Medical Oncology, Heidelberg, Baden-Wurttemberg
  - Technischen Universitat München - Urologische Klinik, München, Bavaria
  - Charité Universitätsmedizin Berlin, Dept. of Interdisciplinary Urology, Berlin
  - Universitätsklinikum Carl Gustav Carus an der Technischen Universität Dresden, Klinik und Poliklinik, Dresden
  - Universitätsklinikum Essen (AöR) Westdeutsches Tumorzentrum, Essen
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum Tübingen, Klinik für Urologie, Tübingen
- Italy (12):
  - Presidio Ospedaliero Antonio Perrino - U.O.C. Oncologia Medica, Brindisi
  - S.C. Oncologia - ASST Cremona P.O. Ospedale di Cremona, Cremona
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Istituto Europeo di Oncologia - Divisione di Oncologia Medica Urogenitale e Cervico Facciale, Milan
  - U.O.C. ASST Santi Paolo e Carlo - Ospedale San Carlo Borromeo, Milan
  - University of Modena and Reggio Emilia (Azienda Ospedaliera-Universitaria Policlinico Modena), Modena
  - Istituto Nazionale Tumori IRCCS "Fondazione G. Pascale", Naples
  - Azienda Ospedaliero Universitaria San Luigi Gonzaga, Orbassano
  - Unità Operativa (UO) di Oncologia Medica - ICS Maugeri, Pavia
  - U.O. Oncologia Ospedale degli Infermi - Dipartimento di Oncologia ed Ematologia, Rimini
  - Policlinico Universitario A. Gemelli, Roma
  - Policlinico Universitario Campus Bio-Medico, Rome
- New Zealand (4):
  - Auckland City Hospital, Auckland, Grafton
  - Christchurch Hospital, Christchurch, South Island
  - Waikato Hospital, Hamilton
  - Wellington Regional Hospital, Wellington
- Spain (13):
  - Hospital Universitario Virgen del Rocío, Seville, Andalusia
  - Hospital Universitari VHIO - Vall d'Hebron Departamento de Oncologia, Barcelona
  - El Hospital Clínic i Provincial de Barcelona (HCPB), Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Institut Català d'Oncologia (ICO) L'Hospitalet, Barcelona
  - Institut Català d'Oncologia, Girona
  - HGU Gregorio Marañon, Madrid
  - MD Anderson Cancer Center Madrid, Madrid
  - El Hospital Universitario 12 de Octubre, Madrid
  - Centro Integral Oncologico Clara Campal (CIOCC) HM, Madrid
  - Hospital Parc Taulí de Sabadell, Sabadell
  - Hospital Universitario Virgen de Macarena, Seville
  - Fundación Instituto Valencia d'Oncología (IVO), Valencia
- United Kingdom (8):
  - The Christie NHS Foundation Trust, Manchester, Greater Manchester
  - Beatson West of Scotland Cancer Centre, Glasgow, Lanarkshire
  - Mount Vernon Cancer Centre, London, Middlesex
  - Nottingham University Hospitals NHS Trust - City Hospital Campus, Nottingham, Nottinghamshire
  - St. Bartholomew's Hospital, Barts Health NHS Trust, London
  - The Royal Marsden NHS Foundation Trust, London
  - Sarah Cannon Research Institute UK Limited, London
  - Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tannir NM, Agarwal N, Porta C, Lawrence NJ, Motzer R, McGregor B, Lee RJ, Jain RK, Davis N, Appleman LJ, Goodman O Jr, Stadler WM, Gandhi S, Geynisman DM, Iacovelli R, Mellado B, Sepulveda Sanchez JM, Figlin R, Powles T, Akella L, Orford K, Escudier B. Efficacy and Safety of Telaglenastat Plus Cabozantinib vs Placebo Plus Cabozantinib in Patients With Advanced Renal Cell Carcinoma: The CANTATA Randomized Clinical Trial. JAMA Oncol. 2022 Oct 1;8(10):1411-1418. doi: 10.1001/jamaoncol.2022.3511. PMID 36048457

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Eligible participants were randomized in a 1:1 ratio to either the Pbo-Cabo arm or the CB-Cabo arm. Randomization was stratified by prior treatment with PD-1/PD-L1 inhibitor therapy (yes vs. no) and the International Metastatic Renal Cell Carcinoma Database Consortium (IMDC) Prognostic Risk Group (favorable vs. intermediate vs. poor).
Groups:
- CB-Cabo: CB-839 800 mg BID + cabozantinib (60 mg once daily [QD]) administered orally on Days 1 through 28 of each 28-day cycle until disease progression per RECIST v1.1 or unacceptable toxicity, whichever occurred first.
Period: Overall Study
Arm/Group | Pbo-Cabo | CB-Cabo
Started | 223 | 221
Received at Least 1 Dose of Study Drug | 221 | 221
Completed (Participants received study treatment until disease progression or unacceptable toxicity, whichever occurred first.) | 0 | 0
Not Completed | 223 | 221
Not completed — Death | 89 | 93
Not completed — Withdrawal by Subject | 8 | 7
Not completed — Lost to Follow-up | 1 | 3
Not completed — Study terminated by sponsor | 124 | 118
Not completed — Other, Not Specified | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pbo-Cabo | CB-Cabo | Total
Number analyzed (Participants) | 223 | 221 | 444
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.7 (10.33) | 60.6 (10.37) | 61.2 (10.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 47 | 115
  Male | 155 | 174 | 329
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 11 | 25
  Not Hispanic or Latino | 173 | 176 | 349
  Unknown or Not Reported | 36 | 34 | 70
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 176 | 174 | 350
  Not Reported | 31 | 32 | 63
  Other, Not Specified | 3 | 9 | 12
  Black or African American | 6 | 3 | 9
  Asian | 6 | 2 | 8
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
Stratification Factor: Prior PD-1/PD-L1 Inhibitor Therapy [Count of Participants; unit: Participants] — PD-1: programmed cell death protein 1 PD-L1: programmed cell death protein ligand 1
  Participants
    Yes | 139 | 137 | 276
    No | 84 | 84 | 168
Stratification Factor: IMDC Category [Count of Participants; unit: Participants] — The International Metastatic renal cell carcinoma Database Consortium (IMDC) score is currently used as prognostic index to stratify patients with mRCC in 3 subgroups: good/favorable, intermediate and poor-risk groups.
  Participants
    Poor | 35 | 35 | 70
    Intermediate | 149 | 147 | 296
    Favorable | 39 | 39 | 78

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) as Assessed by the Independent Radiology Committee (IRC)
Description: PFS is defined as the time from randomization to the occurrence of disease progression as assessed by the IRC using RECIST v1.1 or death from any cause, whichever occurs first. Subjects not experiencing disease progression or death at the time of analysis of PFS will be censored at the date of the last evaluable radiographic disease assessment. RECIST v1.1 criteria:
  Complete Response (CR): Disappearance of all target lesions. Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition, the sum must also demonstrate an absolute increase of at least 5 mm. Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: Up to the primary analysis data cut-off date of 31 Aug 2020. Maximum duration of follow-up for PFS was 22.14 months.
Population: Intent-to-Treat (ITT) Analysis Set: All randomized participants, analyzed according to the treatment group to which they are randomized.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pbo-Cabo | CB-Cabo
Number analyzed (Participants) | 223 | 221
months | 9.33 [7.64 to 11.01] | 9.17 [7.59 to 11.10]
Statistical Analysis 1: Comparison: Pbo-Cabo vs CB-Cabo; Stratified Analysis 1: Stratified by prior programmed cell death protein 1/programmed cell death protein ligand 1 (PD-1/PDL1) inhibitor therapy (yes vs no) and International Metastatic Renal Cell Carcinoma Database (IMDC) prognostic risk group (favorable vs intermediate vs poor); Test type: Superiority; p = 0.6528, Log Rank; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.74 to 1.21]
Statistical Analysis 2: Comparison: Pbo-Cabo vs CB-Cabo; Stratified Analysis 2: Stratified by prior PD-1/PD-L1 inhibitor therapy [yes vs. no] and IMDC prognostic risk group [favorable vs. intermediate/poor]; Test type: Superiority; p = 0.8193, Log Rank; Hazard Ratio (HR) = 0.97, 95% CI 2-sided [0.76 to 1.24]
Statistical Analysis 3: Comparison: Pbo-Cabo vs CB-Cabo; Stratified Analysis 3: Stratified by the number of prior anti-angio cancer therapy [0 vs. >=1]; Test type: Superiority; p = 0.8345, Log Rank; Hazard Ratio (HR) = 0.97, 95% CI 2-sided [0.76 to 1.25]
Statistical Analysis 4: Comparison: Pbo-Cabo vs CB-Cabo; Unstratified Analysis; Test type: Superiority; p = 0.9479, Log Rank; Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.78 to 1.27]

2. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from randomization to death due to any cause. Estimated from Kaplan-Meier methodology. 95% confidence interval (CI) based on Brookmeyer-Crowley methodology.
Time Frame: Up to the primary analysis data cut-off date of 31 Aug 2020. Maximum duration of follow-up for OS was 25.86 months.
Population: ITT Analysis Set: All randomized participants, analyzed according to the treatment group to which they are randomized.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Pbo-Cabo: Placebo BID + cabozantinib (60 mg QD) administered orally on Days 1 through 28 of each 28-day cycle until disease progression per RECIST v1.1 or unacceptable toxicity, whichever occurred first.
Arm/Group | Pbo-Cabo | CB-Cabo
Number analyzed (Participants) | 223 | 221
months | 24.84 [21.59 to NA] — Not estimable due to small number of events. | 22.24 [18.56 to NA] — Not estimable due to small number of events.
Statistical Analysis 1: Comparison: Pbo-Cabo vs CB-Cabo; Stratified Analysis 1: Stratified by prior PD-1/PD-L1 inhibitor therapy [yes vs. no] and IMDC prognostic risk group [favorable vs. intermediate vs. poor]; Test type: Superiority; p = 0.3867, Log Rank; Hazard Ratio (HR) = 1.15, 95% CI 2-sided [0.83 to 1.6]
Statistical Analysis 2: Comparison: Pbo-Cabo vs CB-Cabo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.3367, Log Rank; Hazard Ratio (HR) = 1.17, 95% CI 2-sided [0.85 to 1.62]
Statistical Analysis 3: Comparison: Pbo-Cabo vs CB-Cabo; Stratified Analysis 3: Stratified by prior PD-1/PD-L1 inhibitor therapy [yes vs. no] and IMDC prognostic risk group [favorable vs. intermediate/poor]; Test type: Superiority; p = 0.2416, Log Rank; Hazard Ratio (HR) = 1.22, 95% CI 2-sided [0.88 to 1.69]
Statistical Analysis 4: Comparison: Pbo-Cabo vs CB-Cabo; Unstratified Analysis; Test type: Superiority; p = 0.3043, Log Rank; Hazard Ratio (HR) = 1.19, 95% CI 2-sided [0.86 to 1.64]

3. Secondary Outcome: PFS as Assessed by the Investigator
Description: as for outcome 1
Time Frame: Up to the primary analysis data cut-off date of 31 Aug 2020. Maximum duration of follow-up for PFS was 22.64 months.
Population: ITT Analysis Set: All randomized participants, analyzed according to the treatment group to which they are randomized.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pbo-Cabo | CB-Cabo
Number analyzed (Participants) | 223 | 221
months | 8.38 [6.34 to 9.79] | 9.17 [7.49 to 9.46]
Statistical Analysis 1: Comparison: Pbo-Cabo vs CB-Cabo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.9692, Log Rank; Hazard Ratio (HR) = 1.00, 95% CI 2-sided [0.79 to 1.25]
Statistical Analysis 2: Comparison: Pbo-Cabo vs CB-Cabo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.9235, Log Rank; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.8 to 1.27]
Statistical Analysis 3: Comparison: Pbo-Cabo vs CB-Cabo; Stratified Analysis 3: Stratified by the number of prior anti-angio cancer therapy [0 vs. >=1]; Test type: Superiority; p = 0.9549, Log Rank; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.8 to 1.26]
Statistical Analysis 4: Comparison: Pbo-Cabo vs CB-Cabo; Unstratified Analysis; Test type: Superiority; p = 0.8193, Log Rank; Hazard Ratio (HR) = 1.03, 95% CI 2-sided [0.82 to 1.29]

ADVERSE EVENTS:
Time Frame: All-cause mortality: for a maximum follow-up period of 25.86 months; Intent to Treat Population. Adverse events: From first dose of study drug through at least 28 days after last dose of all study treatments, or until initiation of a new anticancer therapy (if earlier). Overall median duration of safety follow-up was 280.0 days. Safety Analysis Population (all participants who received any study drug, analyzed according to the actual treatment received; 4 Pbo-Cabo participants received CB-Cabo).
Description: Per protocol, Grade 5 disease progression events are excluded from these tables. Disease progression includes events in the preferred terms of disease progression and malignant neoplasm progression.
Arm/Group | Pbo-Cabo | CB-Cabo
All-Cause Mortality (participants affected / at risk) | 89/223 | 93/221
Serious Adverse Events (participants affected / at risk) | 74/217 | 90/225
Other Adverse Events (participants affected / at risk) | 213/217 | 222/225
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pbo-Cabo (N=217) | CB-Cabo (N=225)
Hypertension (Vascular disorders) | 1 | 2
Deep vein thrombosis (Vascular disorders) | 0 | 1
Embolism (Vascular disorders) | 0 | 1
Haemorrhage (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
Thrombophlebitis (Vascular disorders) | 1 | 0
Vena cava thrombosis (Vascular disorders) | 0 | 1
Nerve block (Surgical and medical procedures) | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to pelvis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pregnancy of partner (Social circumstances) | 1 | 0
General physical health deterioration (General disorders) | 2 | 1
Fatigue (General disorders) | 0 | 2
Asthenia (General disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Chills (General disorders) | 0 | 1
Death (General disorders) | 0 | 1
Malaise (General disorders) | 0 | 1
Mucosal inflammation (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 2 | 2
Delirium (Psychiatric disorders) | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 2
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0
Traumatic fracture (Injury, poisoning and procedural complications) | 1 | 0
Troponin I increased (Investigations) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 2
Myocardial infarction (Cardiac disorders) | 1 | 2
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Atrial flutter (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Cardiac ventricular thrombosis (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 7 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 5
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Aphasia (Nervous system disorders) | 1 | 0
Cerebellar syndrome (Nervous system disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Dyskinesia (Nervous system disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Monoplegia (Nervous system disorders) | 0 | 1
Motor dysfunction (Nervous system disorders) | 0 | 1
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 0 | 1
Spinal cord compression (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 6
Vomiting (Gastrointestinal disorders) | 1 | 3
Abdominal pain (Gastrointestinal disorders) | 1 | 2
Ascites (Gastrointestinal disorders) | 0 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 2
Diverticular perforation (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Haemoperitoneum (Gastrointestinal disorders) | 1 | 0
Inguinal hernia strangulated (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Intestinal perforation (Gastrointestinal disorders) | 0 | 1
Melaena (Gastrointestinal disorders) | 1 | 0
Oesophageal food impaction (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Volvulus (Gastrointestinal disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 3 | 1
Hepatitis (Hepatobiliary disorders) | 1 | 1
Bile duct stenosis (Hepatobiliary disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 4 | 2
Haematuria (Renal and urinary disorders) | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 1
Renal colic (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
Urinary bladder haemorrhage (Renal and urinary disorders) | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Fracture pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 2
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1
Pneumonia (Infections and infestations) | 3 | 2
Urinary tract infection (Infections and infestations) | 3 | 1
Appendicitis (Infections and infestations) | 0 | 3
Abscess (Infections and infestations) | 1 | 1
Anal abscess (Infections and infestations) | 1 | 1
Postoperative wound infection (Infections and infestations) | 2 | 0
Tooth infection (Infections and infestations) | 1 | 1
Acute sinusitis (Infections and infestations) | 1 | 0
Appendicitis perforated (Infections and infestations) | 0 | 1
COVID-19 (Infections and infestations) | 0 | 1
COVID-19 pneumonia (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
Cholecystitis infective (Infections and infestations) | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Encephalitis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 0
Joint abscess (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Paraspinal abscess (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 0 | 1
Soft tissue infection (Infections and infestations) | 0 | 1
Wound abscess (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pbo-Cabo (N=217) | CB-Cabo (N=225)
Hypertension (Vascular disorders) | 72 | 82
Hypotension (Vascular disorders) | 13 | 10
Fatigue (General disorders) | 109 | 94
Asthenia (General disorders) | 49 | 49
Mucosal inflammation (General disorders) | 36 | 23
Oedema peripheral (General disorders) | 21 | 22
Pyrexia (General disorders) | 15 | 20
Chest pain (General disorders) | 13 | 9
Insomnia (Psychiatric disorders) | 17 | 21
Anxiety (Psychiatric disorders) | 12 | 16
Depression (Psychiatric disorders) | 16 | 7
Fall (Injury, poisoning and procedural complications) | 12 | 11
Weight decreased (Investigations) | 65 | 77
Alanine aminotransferase increased (Investigations) | 39 | 63
Aspartate aminotransferase increased (Investigations) | 40 | 56
Blood creatinine increased (Investigations) | 12 | 24
Blood alkaline phosphatase increased (Investigations) | 14 | 15
Cough (Respiratory, thoracic and mediastinal disorders) | 41 | 50
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 41 | 33
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 34 | 30
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 16 | 20
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 13 | 21
Anaemia (Blood and lymphatic system disorders) | 29 | 28
Thrombocytopenia (Blood and lymphatic system disorders) | 14 | 20
Dysgeusia (Nervous system disorders) | 52 | 41
Headache (Nervous system disorders) | 32 | 39
Dizziness (Nervous system disorders) | 24 | 23
Paraesthesia (Nervous system disorders) | 12 | 10
Vision blurred (Eye disorders) | 14 | 22
Photophobia (Eye disorders) | 8 | 26
Diarrhoea (Gastrointestinal disorders) | 160 | 162
Nausea (Gastrointestinal disorders) | 118 | 123
Vomiting (Gastrointestinal disorders) | 75 | 77
Constipation (Gastrointestinal disorders) | 63 | 69
Stomatitis (Gastrointestinal disorders) | 49 | 47
Abdominal pain (Gastrointestinal disorders) | 39 | 40
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 24 | 42
Dyspepsia (Gastrointestinal disorders) | 28 | 35
Abdominal pain upper (Gastrointestinal disorders) | 25 | 21
Dry mouth (Gastrointestinal disorders) | 21 | 14
Oral pain (Gastrointestinal disorders) | 15 | 9
Flatulence (Gastrointestinal disorders) | 9 | 14
Proteinuria (Renal and urinary disorders) | 17 | 28
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 87 | 95
Rash (Skin and subcutaneous tissue disorders) | 28 | 40
Pruritus (Skin and subcutaneous tissue disorders) | 20 | 25
Dry skin (Skin and subcutaneous tissue disorders) | 19 | 19
Alopecia (Skin and subcutaneous tissue disorders) | 15 | 16
Hair colour changes (Skin and subcutaneous tissue disorders) | 11 | 20
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 14 | 13
Back pain (Musculoskeletal and connective tissue disorders) | 37 | 43
Arthralgia (Musculoskeletal and connective tissue disorders) | 33 | 33
Pain in extremity (Musculoskeletal and connective tissue disorders) | 27 | 28
Muscle spasms (Musculoskeletal and connective tissue disorders) | 24 | 29
Myalgia (Musculoskeletal and connective tissue disorders) | 19 | 11
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 13 | 14
Muscular weakness (Musculoskeletal and connective tissue disorders) | 9 | 15
Hypothyroidism (Endocrine disorders) | 56 | 66
Decreased appetite (Metabolism and nutrition disorders) | 86 | 83
Hypomagnesaemia (Metabolism and nutrition disorders) | 49 | 48
Hypophosphataemia (Metabolism and nutrition disorders) | 38 | 32
Hypokalaemia (Metabolism and nutrition disorders) | 27 | 25
Hyponatraemia (Metabolism and nutrition disorders) | 30 | 16
Hypocalcaemia (Metabolism and nutrition disorders) | 26 | 18
Hyperkalaemia (Metabolism and nutrition disorders) | 16 | 14
Dehydration (Metabolism and nutrition disorders) | 13 | 15
Hypoalbuminaemia (Metabolism and nutrition disorders) | 14 | 12
Urinary tract infection (Infections and infestations) | 18 | 23
Upper respiratory tract infection (Infections and infestations) | 12 | 20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication by the PI before either a multi-site publication or 18 months after final multi-site study report. PI can only publish their own results and provide 45 days in advance notice. PI must delete any Calithera confidential information from the publication other than study results and give good faith consideration to other comments made by Calithera. The PI must delay the publication for up to 45 days if requested by Calithera and publicly acknowledge Calithera and Pfizer support.

DOCUMENTS (2):
  • Study Protocol (2020-04-09): https://cdn.clinicaltrials.gov/large-docs/17/NCT03428217/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-10): https://cdn.clinicaltrials.gov/large-docs/17/NCT03428217/SAP_001.pdf